CLINICAL TRIAL: NCT02735252
Title: Precision Oncology and Molecular Targeting in Advanced Genitourinary Cancers: Identifying Predictive Markers of Response (The "PROMOTE" Study)
Brief Title: PROMOTE: Identifying Predictive Markers of Response for Genitourinary Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Prostate Cancer Foundation (Other); Strata Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 155518; NCI-2018-02052 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-03-24; First posted 2016-04-12 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Advanced Renal Cell Carcinoma; Advanced Urothelial Carcinoma; Genitourinary Cancer
Keywords: Castration Resistant; Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (10):
- Group A: Androgen Signaling Inhibition (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving treatments that inhibit androgen signaling to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group B: Immunotherapy (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving immunotherapy to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group C: Radiotherapy (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving radiotherapy to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group D: Targeted Therapy Not Otherwise Specified (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving targeted therapy and investigational therapeutics to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group E: DNA Damage Response (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving therapies that target DNA damage response pathways to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group F: Aggressive Variant Disease (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients with variants of disease that display aggressive behavior to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group G1: Castration Sensitive, ADT naïve and ADT < 3 months (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving therapies that target DNA damage response pathways to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group G2:Castration Sensitive,Pre-treated w/ sub-optimal PSA (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving therapies that target DNA damage response pathways to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Group R: Advanced Renal Cell Carcinoma (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving therapies that target DNA damage response pathways to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS
- Cohort U: Advanced Urothelial Carcinoma (Experimental): Tumor biopsies: required prior to treatment and optional at time of disease progression.
  Blood draws: required prior to treatment, every 3 months during treatment, and at time of disease progression.
  Molecular markers will be studied in patients receiving therapies that target DNA damage response pathways to identify predictors of benefit and/or response. Treatments are assigned per investigator discretion.
  Interventions: Other: Systemic therapy; Device: StrataNGS

INTERVENTIONS:
Other: Systemic therapy — Systemic therapy is selected by the physician and is not restricted by the study. Molecular testing will be performed on tissue and blood to identify patterns and relationships with clinical outcomes in each group.
Device: StrataNGS — CLIA-approved assay that is being performed as part of standard of care genomic profiling of patients tumor biopsies. The product currently covers about 90 cancer genes and is able to pick up all the known mutations and other types of genetic alterations across them, he added

SUMMARY:
This is a tissue and blood collection protocol requiring image-guided biopsies of metastatic prostate cancer and other genitourinary malignancies including renal cell carcinoma and urothelial carcinoma. Whenever possible, a new bone lesion or new/progressing soft tissue lesion will be chosen for biopsy as opposed to radiographically stable lesion. Patients will be enrolled in into one of several parallel cohorts based upon disease status or type and the planned systemic therapy following baseline tumor biopsy: (A) Androgen signaling inhibition, (B) Immunotherapy, (C) Radiotherapy, (D) Targeted Therapy/Investigational therapeutic, (E) DNA damage response pathway, (F) Aggressive variant disease, (G1) Castration-sensitive ADT naïve and ADT < 3 months), or (G2) Castration-sensitive pre-treated with sub-optimal PSA nadir >0.2 ng/ml, (R) metastatic renal cell carcinoma and metastatic and (U) urothelial carcinoma.

DETAILED DESCRIPTION:
After performing tumor biopsies and blood collection and processing the biopsies and research blood for comprehensive molecular analysis using established methods for RNA and DNA analysis, we will use Pathway Recognition using Data Integration on Genomic Models (PARADIGM) and Differential Pathway Signature Correlation (DiPSC), computational approaches to pathway activity and predictive signature identification developed at University of California, Santa Cruz. We will also collect blood samples (for circulating tumor DNA, plasma, and serum) and circulating tumor cells from participating patients. Residual paraffin- embedded blocks, frozen tissue, and blood products (serum, plasma, and circulating cells) will be stored in a repository for future testing of candidate predictive markers identified during microarray analysis. We will utilize only Clinical Laboratory Improvement Amendments (CLIA)-certified laboratories(e.g. Strata Oncology) to identify genetic mutations within mCRPC tumors to provide genetic information that can be returned to patient to potentially inform treatment decisions.

Certain genomic sequencing will be performed by Strata Oncology.

Following biopsy and baseline peripheral blood collection, patients will be treated per investigator discretion, with treatment corresponding to assigned patient cohort and initiated within 42 days following baseline tumor biopsy and/or research blood collection. Patients will be evaluated for response to therapy per the standard of care for their specific disease type; such as with monthly serum PSA measurements (may be done at UCSF or at local laboratory) and/or restaging scans (bone scan + CT abdomen/pelvis) (UCSF or local radiology facility). Outcomes on treatment post-biopsy will be recorded, including maximal PSA decline, date of radiographic progression.

At the time of disease progression by Prostate Cancer Working Group 2 (PCWG2) criteria for prostate cancer patients, or by RECIST v1.1 for patients with metastatic renal or urothelial cancer, patients may undergo optional repeat assessment for metastatic tumor biopsy, along with mandatory blood collection for analysis of circulating tumor DNA and circulating tumor cells (CTCs). Following second biopsy at progression, patients should continue to be followed for response to subsequent therapy.

Patients will be followed every 6 months for updates on disease status including post-study therapies and survival status via telephone calls and/or chart review.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed prostate cancer, or other advanced / metastatic genitourinary malignancies for cohorts R (renal cell carcinoma) and U (urothelial carcinoma). Participants without histologically confirmed cancer are eligible if both the treating physician and the study PI agree that the patient's history is unambiguously indicative of advanced prostate cancer (e.g. high Prostate-specific antigen (PSA) responsive to Androgen Deprivation Therapy in prostate cancer)
* Radiographic evidence of metastatic disease amenable to image-guided or excisional biopsy of a metastatic site. Soft-tissue as well as bony metastatic lesions will be considered acceptable. Participants with locally advanced disease only (where the biopsy would be of a prostatic mass) are NOT eligible. Biopsy of newly emerging or progressive metastases is desired and preferable to the biopsy of previously existing stable lesions whenever possible. Patients without lesion amenable to biopsy are still eligible, and have the option of re-assessment for potential of metastatic tumor biopsy upon progression as outlined in the study calendar.
* For participants with metastatic lesion amenable for biopsy:
* Platelets > = 75,000/microliter (μl)
* Prothrombin time (PT) or international normalized ratio (INR) and activated partial thromboplastin time (aPTT) < = 1.5 times the institutional upper limit of normal (ULN) within 14 days prior to biopsy.
* Patients on warfarin, aspirin, or other anti-coagulants are eligible provided they are deemed able to tolerate discontinuation of anti-coagulation prior to the biopsy as per usual standard of care. Conversion to low molecular weight heparin prior to biopsy is permitted per local standard operating procedures, provided there is agreement regarding the procedure between the treating physician, the interventional radiologist and the PI.
* Participants with significant congenital or acquired bleeding disorders (e.g type 3 von Wildebrand's disease, acquired bleeding factor inhibitors) are not eligible.
* Age > 18 yrs
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Ability to understand and the willingness to sign a written informed consent.
* Progression on or following most recent systemic therapy given for:
* Metastatic Renal Cell Carcinoma (RCC) or metastatic urothelial carcinoma (UC) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or for metastatic castration resistant prostate cancer (mCRPC) by Prostate Cancer Working Group 2 (PCWG2) criteria, with progression as defined by one or more of the following:

  1. PSA Progression: PSA level of at least 2 nanograms (ng)/milliliter (ml) which has risen on at least 2 separate measurements, at least one week apart (for prostate cancer participants only)
  2. Disease progression by RECIST v1.1
  3. Bone scan progression: the appearance of >= 2 new lesions (for prostate cancer participants only)
  4. Symptomatic progression in an area of radiologically evident disease
* For prostate cancer participants only, serum testosterone < 50 ng/dL. Participants without prior bilateral orchiectomy are required to remain on Luteinizing hormone-releasing hormone (LHRH) analogue for duration of study. Participants with previously documented denovo primary small cell carcinoma of the prostate are exempt from this criterion. If serum for analysis of testosterone level has been collected but result not available by day of scheduled baseline biopsy, patient may still be eligible for study participation upon at the discretion of the Principal Investigator
* Participants must possess one of the following criteria:

  1. Planned treatment within 42 days following baseline tumor biopsy and/or research blood collection with androgen signaling inhibitor excluding enzalutamide (cohort A), immunotherapy (cohort B), radiotherapy (cohort C), investigational therapeutic (cohort D), or agent targeting the DNA repair pathway including but not limited to platinum chemotherapy or poly adenosine diphosphate-ribose polymerase (PARP) inhibition (cohort E). Therapeutic combinations are allowed and as treatment may fall into more than one category, cohort assignment will be per PI discretion.
  2. Aggressive variant cancer (cohort F), defined by one or more of the following:

     * Presence of one or more visceral organ metastases
     * Serum neuron specific enolase and/or chromogranin A >ULN
     * Progression by PCWG2 criteria within 12 months following initiation of primary androgen deprivation therapy (ADT) +/- chemotherapy for metastatic hormone sensitive prostate cancer
     * Prior histologic evidence of small cell and/or intermediate atypical carcinoma differentiation
* Presence of advanced or metastatic renal cell carcinoma (Cohort R) with planned treatment with a novel agent such as a targeted agent within 42 days following baseline tumor biopsy. Therapeutic combinations are allowed and as treatment may fall into more than one category, cohort assignment will be per PI discretion
* Presence of advanced or metastatic urothelial carcinoma (Cohort U) with planned treatment with a novel agent such as an Antibody Drug Conjugate (ADC) or a targeted agent within 42 days following baseline tumor biopsy. Therapeutic combinations are allowed and as treatment may fall into more than one category, cohort assignment will be per PI discretion.
* Additional inclusion criteria for (cohort G): Metastatic hormone-naïve prostate cancer who are planning to start (Group 1) or currently receiving (Group 2) androgen deprivation therapy. The use of chemotherapy or other investigational agents is allowed but not required in both Group 1 and Group 2.

  * Group 1 (ADT naïve and on ADT < 3 months): Participants who have not received LHRH analogue, LHRH antagonist or any anti-androgen for metastatic disease. Participants who have received ADT in the past 3 months will be included. Prior use of androgen deprivation therapy in the (neo)adjuvant, salvage, or biochemically recurrent setting is allowed provided the last day of effective androgen deprivation was more than 12 months prior to study entry. Androgen deprivation therapy must be planned to start within 28 days of baseline tumor biopsy.
  * Group 2 (ADT Pre-Treated with sub-optimal PSA nadir): Participants who have initiated androgen deprivation therapy (including LHRH agonists, antagonists and/or anti-androgens) for metastatic prostate cancer within 6-12 months prior to study entry who have suboptimal serum PSA nadir > 0.2 ng/mL.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2016-05-25 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of Treatment Benefit by group | Up to 5 years
  Using PARADIGM and DiPSC tools, the investigators will discover genetic expression and clinical factors that are predictive of treatment benefit within each treatment cohort using correlative analysis.
Positive Predictive Value (PPV) | Up to 5 years
  Supervised analysis using response / benefit from the experimental therapy to assess feasibility of pattern recognition/discovery of factors that are associated with response and generate a positive predictive value. Positive predictive value is the probability that participants with a positive test truly have the disease. Positive Predictive Value: True Positive / (True Positive +False Positive)
Median Progression-Free Survival (PFS) | Up to 5 years
  PFS is measured from the time in months of the initiation of therapy after biopsy at enrollment until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or death. For participants initiating treatment, their screening clinical, laboratory, and radiological status will be used as a baseline. Progression is a composite endpoint that can be based upon prostate specific antigen (PSA), objective measures of disease (Response Evaluation Criteria in Solid Tumors (RECIST v.1.1), symptoms, or death.
Median Overall Survival (OS) | Up to 5 years
  OS is measured from the time in months of the initiation of therapy after biopsy at enrollment until death.

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) Response Rate | Up to 5 years
  PSA response rate will be measured as the percentage of change in PSA from baseline to 12 weeks on therapy (or earlier if participants discontinue therapy prior to 12 weeks) as well as the maximum decline in PSA that occurs at any point during treatment
Objective Response Rate (ORR) | Up to 5 years
  ORR is defined as the proportion of participants with a measurable response using either Prostate Specific Working Group 2 (PCWG2) criteria for prostate cancer patients or RECIST v1.1 for genitourinary cancer.
Number of participants with presence of somatic mutations | Up to 5 years
  The presence of somatic mutations (yes/no) in a panel of prostate cancer-related, genitourinary cancer-related and targetable genes will be identified for each participant and will be summarized by mutation using descriptive statistics.
Comparison of pathway activity signatures and overall survival | Up to 5 years
  The log-rank test will be used to test if any identified pathway activity signatures or tumor histologies predicts overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No